CLINICAL TRIAL: NCT01101802
Title: A Prospective, Randomised, Double-blind, Placebo-controlled Trial Evaluating the Effects of Mycophenolate Mofetil on 'Surrogate Markers' for Atherosclerosis in Female Patients With SLE.
Brief Title: Mycophenolate Mofetil in Systemic Lupus Erythematosus (MISSILE)
Acronym: MISSILE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Institute of Child Health, University College London, London, UK. (Unknown)
Responsible Party: Dr David D'Cruz, Lupus Research Unit, St Thomas' hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WX18694; ISRCTN
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2005-05

CONDITIONS: Systemic Lupus Erythematosus; Atherosclerosis
Keywords: SLE; Atherosclerosis; Endothelial function; Mycophenolate mofetil
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Atherosclerosis | interventions — Mycophenolic Acid; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate mofetil (Active Comparator): Patients were given 1gm bd mycophenolate mofetil for 8 weeks
  Interventions: Drug: Mycophenolate mofetil
- Sugar pill (Placebo Comparator)
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Mycophenolate mofetil — Arm 1 patients were given 1 gm bd mycophenolate mofetil for 8 weeks, The mycophenolate was dispensed as 500mg tablets.
  Other Names: Cellcept
  Arms: Mycophenolate mofetil
Drug: sugar pill — Arm 2 patients were given 2 sugar pills bd for 8 weeks
  Arms: Sugar pill

SUMMARY:
Systemic lupus erythematosus (SLE) is an independent risk factor for atherosclerosis. Endothelial dysfunction is the earliest marker of atherosclerosis and is measured by flow mediated dilation (FMD) of the brachial artery. The purpose of the study was to measure FMD in mild, stable SLE patients and look for change in FMD with the immunosuppressant drug mycophenolate mofetil (MMF).

ELIGIBILITY:
Inclusion Criteria:

* Female SLE patients
* Age 18-60 years
* If premenopausal using a reliable method of contraception
* Clinically stable disease
* Taking hydroxychloroquine and up to 15mgs of prednisolone daily

Exclusion Criteria:

* Smokers
* Pregnancy or breast feeding
* Use of other immunosuppressants (hydroxychloroquine and stable dose of prednisolone up to 15 mgs daily will be permitted)
* Use of any investigational drug within 1 month prior to screening
* Acute infections 2 weeks prior to Visit 1
* History of ischaemic heart disease or end stage renal disease
* Current signs or symptoms of severe, progressive or uncontrolled hepatic, haematological, gastroenterological, endocrine, pulmonary, cardiac or neurological disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | 8 weeks
  Measure of endothelial function using doppler ultrasound to measure brachial artery dilation in response to increase blood flow.

SECONDARY OUTCOMES:
BILAG, SLEDAI, | 8 weeks
  Measurements of disease activity in SLE

CONTACTS AND LOCATIONS:
Overall Officials: David P D'Cruz, MD, FRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Lupus Research Unit, St Thomas' Hospital, London, United Kingdom